CLINICAL TRIAL: NCT04171206
Title: A Brief Internet-delivered Intervention to Promote Healthy Relationships Among Young Adults: A Randomised Placebo-controlled Pilot Study
Brief Title: Free From Abuse: The Booster Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sheffield (Other)
Collaborators: University of Huddersfield (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 031298
Record Dates: First submitted 2019-11-13; First posted 2019-11-20 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2019-11

CONDITIONS: Violence, Gender-Based; Violence, Domestic
Keywords: Interpersonal partner violence; Dating violence; Internet-delivered intervention
MeSH Terms: interventions — Technology

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Free From Abuse (Experimental): This is a brief internet-delivered intervention designed to boost participants' ability to recognise abusive behaviour, reduce acceptance of myths related to domestic violence and IPV, as well as decrease abuse perpetration and victimisation.
  Interventions: Other: Free From Abuse
- Technology and crime (Placebo Comparator): This is a brief internet-delivered placebo intervention designed to inform participants about how the development of technology could affect crime.
  Interventions: Other: Technology and crime

INTERVENTIONS:
Other: Free From Abuse — Participants in the treatment arm will watch a 15-minute talk given by an adult female survivor of IPV who tells the story of her abusive relationship. After watching the video, participants will read information on 10 signs of an unhealthy relationship. The intervention will take approximately 25 minutes to complete.
  Arms: Free From Abuse
Other: Technology and crime — Participants in the placebo control arm will watch a 19-minute talk on technology development and crime. After watching the video, participants will read 10 facts about cyber security. The intervention will take approximately 25 minutes to complete.
  Arms: Technology and crime

SUMMARY:
This project is designed to develop and test a brief internet-delivered intervention to promote healthy relationships among young adults.

DETAILED DESCRIPTION:
In spite of the fact that young adults are at an increased risk of experiencing and perpetrating intimate partner violence (IPV), there is a lack of universal and widely accessible prevention programmes targeted at this age group. One of the reasons for this may be that it is difficult to deliver a universal prevention to individuals who are not formally grouped through one organisation, such as employed young adults. Those who are formally grouped, such as university students, are unlikely to take part in a lengthy prevention programme which is not a part of an official curriculum. Therefore, there is a need for widely available, accessible, and efficacious IPV prevention programmes that could be appropriate for all young adults regardless of gender. Since many young adults in contemporary Western societies were exposed to some kind of relationship education in schools, it may be that a brief programme will suffice to further boost their awareness of IPV and reduce IPV perpetration and victimisation risk. Therefore, we propose a brief internet-based intervention, Free From Abuse - The Booster Project, to achieve these objectives.

Primary objectives:

1. To investigate the acceptability and feasibility of the internet-delivered intervention to university students (determined using the 1 and 4-week follow-up rates, % of participants who correctly answered control questions assessing compliance);
2. To assess the acceptability and feasibility of the outcome measures as methods to measure effectiveness of the intervention within a definitive trial (determined using % of missing data);
3. To estimate the standard deviation (SD) for the continuous outcomes to inform sample size calculations for a definitive trial.

Secondary objective:

1. To evaluate the potential effectiveness of the brief internet-delivered intervention, Free From Abuse - The Booster Project, in increasing recognition of abusive behaviour, as well as reducing acceptance of myths about domestic violence, abuse perpetration, and abuse victimisation among young university students compared with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be university students aged between 18-24 years, reside in the UK, have access to a computer and internet connection, and be fluent in English.

Exclusion Criteria:

* Participants will not be eligible to enrol in the trial if they have visual and/or auditory deficits with regards to watching video clips.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 148 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-07-15 (Actual)

PRIMARY OUTCOMES:
Change in recognition of abusive behaviour | baseline, immediately post intervention - an average of 1 hour, 1 week, 4 weeks
  Recognition of adolescent relationship abuse (ARA) scale (Rothman, Decker, & Silverman, 2006); scores on this 12-item self-report scale range from 12 to 60, with higher scores indicating an increased recognition of abusive behaviour
Change in acceptance of myths about domestic violence | baseline, immediately post intervention - an average of 1 hour, 1 week, 4 weeks
  Domestic Violence Myth Acceptance Scale (DVMAS; Peters, 2008); scores on this 18-item self-report scale range from 18 to 108, with higher scores indicating an increased acceptance of myths about domestic violence

SECONDARY OUTCOMES:
Change in abuse perpetration | baseline, 4 weeks
  Safe Dates - Psychological Abuse Perpetration scale (Foshee et al., 1996, 1998); scores on this 14-item self-report scale range from 14 to 56, with higher scores indicating an increased abuse perpetration
Change in abuse victimisation | baseline, 4 weeks
  14-item Safe Dates - Psychological Abuse Victimisation scale (Foshee et al., 1996, 1998); scores on this 14-item self-report scale range from 14 to 56, with higher scores indicating an increased abuse victimisation

CONTACTS AND LOCATIONS:
Overall Officials: Agata Debowska, PhD, Principal Investigator — University of Sheffield
Locations (1):
- The University of Sheffield, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: No